CLINICAL TRIAL: NCT00877357
Title: Open Label Multicentric Randomized Phase IV Post Marketing Safety, Immunogenicity and Lot-to-Lot Consistency Analysis of Shan 5 [DTPwHB-Hib (Liquid) Pentavalent Combination Vaccine] in Indian Infants
Brief Title: Safety, Long Term Immunogenicity and Lot Consistency Study of Liquid Pentavalent Combination Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shantha Biotechnics Limited (Industry)
Responsible Party: VP, Scientific and Medical Affairs, Shantha Biotechnics Limited
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SBL/DTPwHBHib/WHOCON/2008/0100
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-04

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Haemophilus Influenzae Type B
Keywords: Vaccine; Prevention; Diphtheria; Tetanus; Pertussis; Hepatitis B; Haemophilus influenzae type b; Lot Consistency; Long Term Immunogenicity; Reactogenicity; Healthy infants
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Haemophilus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Shan 5 Lot No 1 (Experimental)
  Interventions: Biological: Shan 5
- Shan 5 Lot No 2 (Experimental)
  Interventions: Biological: Shan 5
- Shan 5 Lot No 3 (Experimental)
  Interventions: Biological: Shan 5

INTERVENTIONS:
Biological: Shan 5 — Diphtheria, tetanus, whole cell pertussis, recombinant hepatitis B and Hib tetanus toxoid conjugate pentavalent liquid combination vaccine

SUMMARY:
A randomized phase IV study of the liquid pentavalent combination vaccine to evaluate the safety, immunogenicity (short term and long term) and clinical consistency of three production lots of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children in the age group six to eight weeks
* Born after a normal gestational period (36 - 42 weeks)
* Mother's HBsAg (hepatitis B surface antigen) assured negative.
* Father, mother or legally acceptable representative properly informed about the study and having signed the informed consent form.

Exclusion Criteria:

* Administration of immunoglobulin or any blood products since birth.
* Use of any investigational, un-registered drug, or vaccine other than the study vaccine (with the exception of oral polio vaccination OPV & BCG vaccine) during the study period or within 30 days preceding the first dose of the study vaccine.
* Previous vaccination or evidence of infection with DTP or Hib.
* History of allergic disease or reaction likely to be exacerbated by any component of the vaccine including allergy to antibiotics.
* Major congenital or hereditary immunodeficiency.
* Infants born to mothers known to be HIV positive.
* Infants having evidence of disease or fever, history of allergic disease or persistent hematological, hepatic, renal, cardiac or respiratory disease and signs of a CNS disorder at the time of vaccination.
* Infants showing any of the following reactions after any dose of study vaccine will be withdrawn for subsequent doses: body temperature more than 40.40C, persistent screaming or crying for 3 hours within 48 hours of vaccination, seizures, encephalopathy and hypersensitivity reaction.
* Parent/s or guardian of subject unable to maintain diary card

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Solicited and unsolicited local and systemic adverse events following vaccination | 4 Months

SECONDARY OUTCOMES:
Seroprotection rates for Diphtheria, Tetanus, Pertussis, Hepatitis B and Hib following 3 doses of the vaccine | 12 Months
Lot Consistency based on safety and Seroprotection rates for Diphtheria, Tetanus, Pertussis, Hepatitis B and Hib following 3 doses of the vaccine from each of the three lots | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Raman Rao, MD, Study Director — Shantha Biotechnics Limited
Locations (1):
- School of Public Health, Post Graduate Institute of Medical Education and Research, Chandigarh, Uttarakhand, India